CLINICAL TRIAL: NCT05843110
Title: Decision-making Process of Couples Confronted With Prenatal Diagnosis of an Isolated CCA
Acronym: ACCED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP 200309
Record Dates: First submitted 2022-02-09; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-02

CONDITIONS: Corpus Callosum Agenesis
Keywords: Corpus callosum agenesis; pregnancy; decision
MeSH Terms: conditions — Agenesis of Corpus Callosum

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision-making process (Other): 1 arm with 25 couples who had an isolated CCA announcement during pregnancy and who decided to continue the pregnancy and 25 couples who had an isolated CCA announcement during pregnancy and who decided to terminate the pregnancy
  Interventions: Other: Decision-making process

INTERVENTIONS:
Other: Decision-making process — Retrospective evaluation using scales, questionnaires and a semi-structured interview

SUMMARY:
This research promoted by the AP-HP (DRCI) is financed by the Agence de la biomédecine (ABM) and the Fondation Maladie Rare (FMR) and received a favourable opinion from the CPP on 8/12/2020. It aims to describe the decision-making process of couples faced with the discovery of an isolated corpus callosum anomaly in their fetus during pregnancy. Indeed, the anomaly of the corpus callosum in antenatal represents a paradigmatic situation of the clinic of uncertainty for couples and teams, because the prognosis is variable, in 80% of the cases it is favourable and in 20% it is associated with an intellectual deficiency. This study will use a mixed methodology, combining quantitative data (STAI A and B anxiety scale, BDI-II depression scale, PCL-5 post-traumatic stress scale, DAS-16 marital relationship dynamics scale, experimental emotional self-evaluation scales adapted to each member of the couple, R/S scale) and qualitative data (through a research interview of the couple conducted by a research psychologist). In the course of the study, 50 couples will be interviewed between 3 months and 5 years after the pregnancy (post-medical termination of pregnancy and post-delivery), with 25 couples who will have continued the pregnancy and 25 couples who will have terminated the pregnancy. Statistical and qualitative analysis of the data using NVivo software will be performed. The aim is to better understand the factors that lead couples to decide to continue or terminate a pregnancy in a situation of extreme prognostic uncertainty, their experience of their decision and to improve the care pathway currently offered to these couples faced with this type of situation.

DETAILED DESCRIPTION:
Couples facing with the discovery of fetal isolated CCA during pregnancy find themselves in a paradigmatic situation of decision-making in a context of extreme uncertainty. They must decide whether to continue or to terminate the pregnancy based on statistical probabilities regarding neurodevelopmental prognosis: favourable in about 80% of cases and associated with an intellectual disability (ID) in about 20% of cases, of variable severity (5% severe). This complex decision belongs to each couple. In situations of prenatal diagnosis it is currently known that the predominant factors in decision-making are related to medical information and to subjective parental perception of the consequences of this information (the potential suffering of the child, the impact on family life, the quality of life of the child, etc.). Prognosis' uncertainty complicates this decision-making and brings couples into significant distress which they express in consultation.

How do couples make their decision? How do they experience this decision over time? These questions have not yet been the subject of a specific study concerning decision-making in a context of an uncertain prognosis. It seems essential to better identify the decision-making mechanisms at stake and to understand the experience of this decision-making over time. Findings of this study could improve current practices in support of concerned couples.

More broadly, given the global development of technological advances in prenatal diagnosis (particularly in imaging and genetics), couples are and will increasingly be facing situations of high prognostic uncertainty. A better understanding of the decision-making process concerning the outcome of pregnancy seems essential, as well as the psychological impact of this decision - whatever it may be - on couples. The conclusions of this study, focused on a paradigmatic situation, could be applied to others. Rooted in an interdisciplinary approach, it is crucial that the teams question their practice to improve couples' support during and after pregnancy in all disciplines involved. Finally, technological progress leads to questions that raise ethical and societal issues. This study may provide possible methods ways of response. The main objective of this research is to study the conscious and unconscious factors involved in the couples' decision-making process regarding the outcome of pregnancy in the context of prenatal diagnosis of isolated CCA. Moreover, the investigators aim to study the couples' experiences concerning their decision to continue or terminate the pregnancy and the psychological impact of this decision. The investigators want to evaluate the impact of time on the experience of their decision. The investigators expect to identify the needs of the people involved in order to re-evaluate the practices and improve the care pathway currently proposed.

The study population includes couples who had a fetal announcement of isolated CCA during pregnancy. Both members are 18 years of age or older benefiting from the social security system. They will be included in the study from 3 months to 5 years after the end of the pregnancy (delivery or termination). Signed informed and free consent for each individual is obtained.

Couples for whom a new pregnancy is in progress, one of whose members does not speak French and/or is under legal protection and/or is under a security measure and/or suffers from a decompensated psychiatric pathology known at the time of recruitment cannot be included.

Two groups (50 couples recruited) will be formed in the following way: a first group of 25 couples, who had announcement of fetal isolated CCA during the pregnancy and decided to continue the pregnancy; a second group of 25 couples, who had an announcement of fetal isolated CCA during the pregnancy and decided to terminate the pregnancy.

To address the study objectives, this study uses mixed methods:

The experimental adapted emotional self-evaluation scales (R/S scales). The investigators use retrospective choice self-assessment scales that measure the emotional state associated with the decision and the desire to modify/reconsider the initial choice ("regret" or "relief" gradient). The terms of these scales were adapted in collaboration with Sylvain Moutier to fit the research context, based on our clinical experience.

Anxiety scales (STAI A and B). The STAI inventory is one of the most widely used anxiety assessment scales. Validated in French, it is composed of 40 items that evaluate trait anxiety (the subject's usual anxious temperament) and state anxiety (current anxiety at the time of the interview). The evaluation of these two levels of anxiety and the data already available for the general population constitute the major interest of this scale.

A depression scale: Beck Depression Inventory (BDI-II). This is an inventory measuring the depth of depression. This scale is designed to measure the subjective aspects of depression. It is one of the most widely used scales for the subjective measurement of depression as a complement to clinical investigation. Because of its brevity, BDI-II is well accepted by patients and easy to administer.

The post-traumatic stress disorder Checklist version DSM-5 (PCL-5). This scale is used to assess the state of post-traumatic stress disorder. It measures the three main subsyndromes of PTSD: re-experiencing, avoidance, hypervigilance. Participants graduate their symptoms based on the last month prior to taking the scale.

The revised Dyadic Adjustment Scale-16 (DAS-16) inventory. This is an abridged and revised version of the Dyadic Adjustment Scale (DAS). It studies a couple's reciprocal dyadic adjustment, which would be evolutionary: thus, it measures each partner's overall perception of their conjugality and possible marital distress.

Finally, there is a semi-structured research interview. An interview guide was developped which was submitted to the members participating in the development of this research, during the meetings of the steering committee (COPIL). This interview allows us to study the following elements: account and scope of the abnormality's announcement; their experiences of various specialists' discourses ; content and scope of the information received (probabilities, multitude of scenarios possible....); how can evolve their representations of their baby ; the pregnancy's experience ; anticipation or difficulty in anticipating the consequences of the final decision in relation to uncertainty and doubt; how such a decision may or may not be made by two people; the opinion of others (family, friends, doctors...). This interview is based on the long experience of the investigators in supporting concerned couples. The choice for using a semi-structured research interview was made for several reasons. First, it allows having varied contents and themes specific to every participant. Within each theme, it enables studying the thought process and having information on the effects. It is also a valuable tool in accessing the subjective information of the subject. When used with couples, it allows studying couple dynamics.

Through these scales and interview, the following hypotheses are tested. Firstly, it is assume that the psychological impact of decision making following the announcement of fetal isolated CCA is correlated with decision making (G1: continuation of pregnancy and G2: IMG).

The investigators also believe that in couples who continued the pregnancy (G1), the psychological impact of decision making is correlated to the subjective parental perception of their child's degree of impairment.

Finally, the pre-existing representations of disability in general are considered; the subjective risk of disability related to isolated CCA; pregnancy history; family support; marital alliance, and medical discourse and attitudes facilitated or hindered the couple's decision-making.

Couples (who have been followed since 2017) will be informed of the research during a consultation as part of their routine care (post-MIG consultation, child follow-up consultation, etc.) by one of the physicians or midwives participating in the study at one of the 3 participating centers (Neuropediatrics Department, Armand Trousseau Hospital, Fetal Medicine Department, Armand Trousseau Hospital and Genetics Department, Pitié-Salpêtrière Hospital).

The physician in charge of this consultation during which he informs couples of the research and gives them the study information. They are given a one-week period of reflection and a telephone call will be made by the psychologist-researchers to find out the couple's response (whether they wish to participate or not in this study).

If the couple agrees to participate in the study, an appointment is scheduled at the recruiting center (genetics department) with a psychologist-researcher (associate investigator). During this visit, the investigator (psychologist-researcher) takes time with the two members of the couple to present the study again (taking over the information note given by the doctor) and to answer any questions they may have. The research psychologist checks inclusion and non-inclusion criteria and then collect the free, informed, written consent of each member of the couple. Then, each member of the couple completes the first part of the experimental adapted emotional self-evaluation scales (R/S scales), the anxiety scales (STAI A and B), the depression scale (BDI-II), the post-traumatic stress disorder scale (PCL-5) and the revised inventory of the dyadic adjustment scale (DAS-16). The semi-structured research interview is conducted with the two couple members present. Finally, the second phase of the experimental adapted emotional self-assessment scales (R/S scales) is completed. It is assumed that the appointment may last nearly 3 hours.

The benefits for the couples who agree to participate in this study could be meeting with the psychologist-researchers, i.e. to have time to be heard and to elaborate their experience. The post-pregnancy consultations (in neuropediatrics and genetics) show that couples wish to talk about pregnancy and their choices. Participation in this study may have positive psychological effects. For example: meeting professionals who have clinical experience in accompanying couples in an antenatal diagnosis, a feeling of not being alone, being able to contribute to the improvement of the care pathway for the future couples involved. There is no medical benefit to participating in this research.

Any major risk for the couples invited to participate in this study have not been forcast. However, the research information letter, the scales and the interview may reactivate painful effects. The investigators anticipate that anyone who has received information about this research, whether they participate or not will have the opportunity to be referred to a psychologist if they so desire.

This research promoted by the AP-HP (DRCI) is funded by the Agence de la biomédecine (ABM) and the Rare Disease Foundation (FMR) and has received a positive opinion from the CPP on 8/12/2020.

ELIGIBILITY:
Inclusion Criteria:

1. Couples of which the 2 members are aged 18 and over
2. Couples who have been notified of a fetal isolated CCA
3. Inclusion in the study 3 months to 5 years after the end of pregnancy (delivery or IMG)
4. Collection of free, informed and written consent from each of the 2 members of the couple for their participation in research
5. 2 members of the couple beneficiaries of a social security scheme (beneficiary or entitled outside AME)

Exclusion Criteria:

1. Couples of which one member does not speak French
2. Couples in which one of the members suffers from a decompensated psychiatric pathology known at the time of recruitment
3. Couples for whom a new pregnancy is in progress
4. Couples in which one of the members is under legal protection measure or under security measure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-10-22 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
By using an inductive methodology, the factors (conscious and unconscious) involved in decision-making in couples regarding the outcome of pregnancy in the context of prenatal isolated CCA diagnosis will be determinated. | During the one research interview at the inclusion visit
  Explored in the interview :
  * The development of the child perceived by the parents
  * The subjective risk of disability linked to an isolated CCA
  * Representations of disability in general, preexisting in pregnancy
  * The history of pregnancy before the discovery of the fetal abnormality: experience of the pregnancy since its confirmation and until the discovery of the anomaly, perceptions and representations around the fetus-baby, positive or negative events concerning pregnancy
  * Family support: do couples feel supported by their families? did they perceive an agreement or disagreement as to their decision
  * Discourse and medical attitudes perceived by couples towards the possibilities of TOP or prosecution The interviews are audio registered and fully transcripted. Afterwards they will be analysed through a thematic analysis, in support of NVivo Software. This metodology will give access to qualitative and quantitive datas of the interview.

SECONDARY OUTCOMES:
Study the traumatic impact of the decision | This secondary outcome will be assess at the inclusion visit
  The traumatic impact will be assess through the score on the PCL-5 scale
Evaluate the anxiety within the couples of the study | This other outcome will be assess at the inclusion visit
  Anxiety will be assess through the STAI score
Evaluate the depression within the couples of the study | This other outcome will be assess at the inclusion visit
  Depression will be assess through the BDI-II score
Evaluate the conjugal factors | This other outcome will be assess at the inclusion visit
  The level of conjugal harmony will be assess through the DAS-16 score
Evaluate the degree of confidence in the decision | This other outcome will be assess at the inclusion visit
  The level of regret versus relief will be asses through the score on the R / S scales
Describe the needs of the couples | This other outcome will be assess at the inclusion visit
  It will be assess through the qualtitative analyse of the interview, using Nvivo software " It will be assess through the qualtitative analyse of the interview, using Nvivo software

CONTACTS AND LOCATIONS:
Overall Officials: Delphine HERON, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié-Salpêtrière Hospital, AP-HP - Department of Medical Genetics, Paris, France

IPD SHARING:
Plan to Share IPD: No